CLINICAL TRIAL: NCT04618367
Title: HAIC Combined With Lenvatinib and Sintilimab for Hepatocellular Carcinoma With Portal Vein Tumor Thrombus
Brief Title: HAIC Combined With Lenvatinib and Sintilimab for Hepatocellular Carcinoma With PVTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Zhou Qunfang, MD, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GYEYJR-1
Record Dates: First submitted 2020-10-31; First posted 2020-11-05 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Carcinoma, Hepatocellular; Liver Neoplasms; Sintilimab; Portal Vein Tumor Thrombus
Keywords: Carcinoma, Hepatocellular; lenvatinib; Sintilimab; portal vein tumor thrombus; oxaliplatin; 5-fluorouracil; leucovorin
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — lenvatinib; sintilimab; Antibodies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HAIC plus Lenvatinib and Sintilimab (Experimental): Hepatic arterial infusion of oxaliplatin , fluorouracil, and leucovorin every 6 weeks. Lenvatinib 12 mg (or 8 mg) once daily (QD) oral dosing. Toripalimab 200 mg intravenously every 3 weeks.
  Interventions: Procedure: Hepatic arterial infusion chemotherapy; Drug: Lenvatinib; Drug: Sintilimab

INTERVENTIONS:
Procedure: Hepatic arterial infusion chemotherapy — administration of oxaliplatin , fluorouracil, and leucovorin via the tumor feeding arteries every 6 weeks
Drug: Lenvatinib — 12 mg (or 8 mg) once daily (QD) oral dosing.
  Other Names: TKI inhibits
Drug: Sintilimab — 200mg intravenously every 3weeks
  Other Names: programmed cell death protein-1 (PD-1) antibody

SUMMARY:
This study intends to evaluate the efficacy and safety of hepatic arterial infusion chemotherapy of oxaliplatin, 5-fluorouracil and leucovorin plus lenvatinib and Sintilimab for patients hepatocellular carcinoma and portal vein tumor thrombus.

DETAILED DESCRIPTION:
Hepatic arterial infusion chemotherapy (HAIC) of oxaliplatin, 5-fluorouracil and leucovorin was effective and safe for hepatocellular carcinoma. Lenvatinib was non-inferior to sorafenib in overall survival in untreated advanced hepatocellular carcinoma, and Sintilimab, an programmed cell death protein-1 (PD-1) antibody, was effective and tolerable in patients with hepatocellular carcinoma and portal vein tumor thrombus. No study has evaluated HAIC plus Lenvatinib and Sintilimab. Thus, the investigators carried out this prospective, single-arm study to find out it.

ELIGIBILITY:
Inclusion Criteria:

* 1. clinical diagnosis of HCC; 2. age between18 and 75 years; 3. refused to sorafenib treatment; 4. type I PVTT, type II PVTT, or type III PVTT. 5. Child-Pugh class A or B; 6. Eastern Cooperative Group performance status (ECOG) score of 0-2; 7. Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/L Serum albumin ≥ 32 g/L ASL and AST ≤ 5 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3 8. Prothrombin time ≤18s or international normalized ratio < 1.7. 9. Ability to understand the protocol and to agree to and sign a written informed consent document.

Exclusion Criteria:

* 1. Diffuse HCC; 2. Extrahepatic metastasis; 3. Obstructive PVTT involving both the left and right portal vein or main portal vein.

  4. Serious medical comorbidities. 5. Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy 6. Known history of HIV 7. History of organ allograft 8. Known or suspected allergy to the investigational agents or any agent given in association with this trial.

  9. Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy 10. Evidence of bleeding diathesis. 11. Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Progression free survival rate at 6 months | 6 months
  Progression was defined as progressive disease by independent radiologic review according to mRECIST or death from any cause

SECONDARY OUTCOMES:
Overall survival (OS) | 6 months
  OS is the length of time from the date of randomization until death from any cause.
Progression free survival (PFS) | 6 months
  PFS is defined as the time from the date of randomization to the date of the first objectively documented tumor progression or death due to any cause.
Objective response rate (ORR) | 6 months
  ORR, as determined based on tumor response according to RECIST 1.1, is defined as the proportion of all randomized subjects whose best overall response (BOR) is either a CR or PR.
Adverse events | 6 months
  Safety will be evaluated according to the NCI CTCAE Version 4.03. All observations pertinent to the safety of the study medication will be recorded on the CRF and included in the final report.

CONTACTS AND LOCATIONS:
Overall Officials: Kangshun Zhu, MD, Study Director — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No